CLINICAL TRIAL: NCT07205029
Title: "Predictive Models of Human Body Morphological Evolution to Improve Adherence and Motivation in Dietary-Nutritional Treatments for Overweight and Obesity" [Modelos Predictivos de la Evolución Morfológica Del Cuerpo Humano Para Mejorar la Adherencia y Motivación en Tratamientos Dietético-nutricionales Del Sobrepeso y la Obesidad].
Brief Title: "Predictive Models of the Morphological Evolution of the Human Body to Improve Adherence and Motivation in Dietetic-nutritional Treatments of Overweight and Obesity" [Modelos Predictivos de Evolución Corporal Para Mejorar la Adherencia en Tratamientos de Sobrepeso y Obesidad]
Acronym: Tech4D-Predict
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jorge Azorin Lopez (Other)
Collaborators: Instituto de Investigación Sanitaria y Biomédica de Alicante (Network)
Responsible Party: Sponsor-Investigator, Jorge Azorin Lopez, Principal Investigator. Full professor at the University of Alicante., University of Alicante
Organization: University of Alicante (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UA-2021-11-18; PID2023-149562OB-I00 (Other Grant/Funding Number: Ministerio de Ciencia e Innovación y Universidades. Gobierno de España (MICIU/AEI/10.13039/501100011033 y FEDER/UE). [M)
Record Dates: First submitted 2025-09-18; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Body Image; Executive Function (Cognition); Obesity &Amp;Amp;Amp; Overweight
Keywords: obesity treatment; Virtual Reality intervention; Executive function in overweight and obese individuals; Body image perception; 4D model
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Over a 6-month period, the control group received nutritional recommendations based on the Mediterranean Diet from the nutritionist. In each session, the participant went through the 4D modelling machine, which captures the morphological changes of each individual over time. The control group did not visualise these morphological changes through the virtual reality goggles. Personal and sociodemographic data, clinical information, general health status, anthropometric, nutritional, and lifestyle data, as well as psychological and neuropsychological variables, were collected at two time points: at the beginning (pre-test measures) and at the end of the intervention (post-test measures).
  Interventions: Combination Product: Control: Nutritional intervention
- Experimental group (Experimental): Over a 6-month period, the experimental group received nutritional recommendations based on the Mediterranean Diet from the nutritionist. In each session, the participant went through the 4D body modelling machine, which captures the morphological changes of each participant over time. The experimental group observed the changes in their bodies through immersive virtual reality goggles. After visualising their bodies, all participants in the experimental group completed a questionnaire designed to assess their perception of body image. Personal and sociodemographic data, clinical information, general health status, anthropometric, nutritional, and lifestyle data, as well as psychological and neuropsychological variables, were collected at two time points: at the beginning (pre-test measures) and at the end of the intervention (post-test measures).
  Interventions: Combination Product: Experimental: Nutritional and Virtual reality intervention

INTERVENTIONS:
Combination Product: Experimental: Nutritional and Virtual reality intervention — Over a 6-month period, the experimental group received nutritional recommendations based on the Mediterranean Diet from the nutritionist. In each session, the participant went through the 4D body modelling machine, which captures the morphological changes of each participant over time. The experimental group observed the changes in their bodies through immersive virtual reality goggles. After visualising their bodies, all participants in the experimental group completed a questionnaire designed to assess their perception of body image. Personal and sociodemographic data, clinical information, general health status, anthropometric, nutritional, and lifestyle data, as well as psychological and neuropsychological variables, were collected at two time points: at the beginning (pre-test measures) and at the end of the intervention (post-test measures).
  Arms: Experimental group
Combination Product: Control: Nutritional intervention — Over a 6-month period, the control group received nutritional recommendations based on the Mediterranean Diet from the nutritionist. In each session, the participant went through the 4D modelling machine, which captures the morphological changes of each individual over time. The control group did not visualise these morphological changes through the virtual reality goggles. Personal and sociodemographic data, clinical information, general health status, anthropometric, nutritional, and lifestyle data, as well as psychological and neuropsychological variables, were collected at two time points: at the beginning (pre-test measures) and at the end of the intervention (post-test measures).
  Arms: Control group

SUMMARY:
The objective of this clinical trial is to evaluate the effect of a personalized intervention based on the benefits of 4D body modeling and virtual reality techniques, combined with a dietary-nutritional treatment focused on the Mediterranean Diet, as a tool to improve motivation for change, adherence to treatment and health parameters in patients with overweight and obesity. The main research questions to be addressed are:

* How can a 4D computer vision model combined with virtual reality improve clinical diagnoses, the analysis of morphological changes in the human body over time, and adherence to dietary-nutritional treatment?
* Does adherence to an intensive multifactorial dietary-nutritional treatment based on the Mediterranean Diet (MD), supported by 4D immersive virtual reality technology, lead to improvements in cognitive functioning?
* What impact does a nutritional intervention program based on the Mediterranean Diet and the use of virtual reality have on body image perception?
* Can an intensive intervention based on the Mediterranean Diet and 4D virtual reality technology improve overall health? Researchers will compare the control group (which will receive nutritional recommendations based on the Mediterranean Diet) with the experimental group (which will receive nutritional recommendations based on the Mediterranean Diet and visualize their morphological changes through VR) to determine whether a personalized intervention based on the benefits of 4D modeling and virtual reality, combined with a Mediterranean Diet-focused treatment, is effective in addressing overweight and obesity.

Participants are expected to:

* Follow the dietary-nutritional recommendations throughout the 6-month intervention.
* Visit the clinic once a month for follow-up.
* Complete all clinical and psychological assessments.

ELIGIBILITY:
Inclusion Criteria:

* a BMI greater than 24.9 kg/m2 [overweight (25 ≥ BMI < 30) and obese (BMI ≥ 30)] according to the BMI classification of the WHO;
* the ability to read and write fluently;
* Spanish as a mother tongue.

Exclusion Criteria:

* currently being or having been in dietetic-nutritional treatment supervised by a nutritionist in the last year;
* the presence of an endocrine-metabolic disorder (including thyroid, pituitary gland, and adrenal gland problems and metabolic syndrome);
* the presence of a previous history of neurological disease (e.g., stroke or Parkinson's disease) or a history of head trauma;
* the presence of a history of severe psychopathology according to the diagnostic criteria of the DSM-IV-TR;
* currently receiving psychiatric treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | From enrollment to the end of treatment at 6 months
  BMI was calculated as weight (kg) divided by height squared (m²). According to the WHO classification, overweight will be defined as a BMI ≥ 25.0 kg/m² and obesity as a BMI ≥ 30.0 kg/m².
Weight | From enrollment to the end of treatment at 6 months.
  Body weight (kg) measured using a calibrated digital scale, a TANITA MC-780MA P digital scale (TANITA Corporation, Arlington Heights, IL, USA). Unit of Measure: kilograms (kg).
Height | From enrollment to the end of treatment at 6 months
  Height measured in standing position without shoes using a SECA 213 portable stadiometer (SECA, Hamburg, Germany). Unit of Measure: meters (m)
Body fat | From enrollment to the end of treatment at 6 months
  Body fat percentage measured using a TANITA MC-780MA P digital scale (TANITA Corporation, Arlington Heights, IL, USA). Unit of Measure: percent (%)
Visceral fat | From enrollment to the end of treatment at 6 months
  Visceral fat percentage measured using the TANITA MC-780MA P digital scale. Unit of Measure: percent (%).
Trunk fat | From enrollment to the end of treatment at 6 months
  Fat percentage in the trunk region measured using the TANITA MC-780MA P digital scale. Unit of Measure: percent (%).
Fat in Right Arm | From enrollment to the end of treatment at 6 months
  Fat percentage in the right arm measured using the TANITA MC-780MA P digital scale. Unit of Measure: percent (%).
Fat in Left Arm | From enrollment to the end of treatment at 6 months
  Fat percentage in the left arm measured using the TANITA MC-780MA P digital scale. Unit of Measure: percent (%).
Fat in Right Leg | From enrollment to the end of treatment at 6 months
  Fat percentage in the right leg measured using the TANITA MC-780MA P digital scale. Unit of Measure: percent (%).
Fat in Left Leg | From enrollment to the end of treatment at 6 months
  Fat percentage in the left leg measured using the TANITA MC-780MA P digital scale. Unit of Measure: percent (%).
Waist Circumference | From enrollment to the end of treatment at 6 months
  Waist measured with a flexible measuring tape with 0.1 cm precision. Measurements performed twice. Unit of Measure: centimeters (cm).
Hip Circumference | From enrollment to the end of treatment at 6 months
  Hip measured with a flexible measuring tape with 0.1 cm precision. Measurements performed twice. Unit of Measure: centimeters (cm).
Waist-Hip Ratio (WHR) | From enrollment to the end of treatment at 6 months
  Calculated as the ratio of waist to hip circumference. Unit of Measure: ratio (unitless).
Wrist Circumference | From enrollment to the end of treatment at 6 months
  Measured using a flexible measuring tape with 0.1 cm precision. Measurements performed twice. Unit of Measure: centimeters (cm).
Muscle Mass | From enrollment to the end of treatment at 6 months
  Total body muscle mass measured using the TANITA MC-780MA P digital scale. Unit of Measure: kilograms (kg).
Total Body Water | From enrollment to the end of treatment at 6 months
  Total body water percentage measured using the TANITA MC-780MA P digital scale. Unit of Measure: percent (%).
Glucose Level | From enrollment to the end of treatment at 6 months.
  Capillary glucose measured using the Accutrend® Plus device (Roche Diagnostics GmbH, Mannheim, Germany) from 15-40 μL blood collected via finger prick (Accu-Chek® Softclix® Pro lancing device). Unit of Measure: mg/dL
Total Cholesterol | From enrollment to the end of treatment at 6 months.
  Capillary total cholesterol measured using the Accutrend® Plus device (Roche Diagnostics GmbH, Mannheim, Germany) from 15-40 μL blood collected via finger prick (Accu-Chek® Softclix® Pro lancing device). Unit of Measure: mg/dL
Triglycerides | From enrollment to the end of treatment at 6 months.
  Capillary triglycerides measured using the Accutrend® Plus device (Roche Diagnostics GmbH, Mannheim, Germany) from 15-40 μL blood collected via finger prick (Accu-Chek® Softclix® Pro lancing device). Unit of Measure: mg/dL
Systolic Blood Pressure | From enrollment to the end of treatment at 6 months.
  Measured using the M7 Intelli IT sphygmomanometer (OMRON, M7, Corp., Kyoto, Japan). Unit of Measure: mmHg.
Diastolic Blood Pressure | From enrollment to the end of treatment at 6 months.
  Measured using the M7 Intelli IT sphygmomanometer (OMRON, M7, Corp., Kyoto, Japan). Unit of Measure: mmHg.
Interleukin 6 (IL-6) | From enrollment to the end of treatment at 6 months.
  IL-6 measured from peripheral blood obtained via venipuncture using a bead-based multiplex assay (xMAP) with Luminex 200 flow cytometer. Unit of Measure: pg/mL.
Tumor Necrosis Factor Alpha (TNF-α) | From enrollment to the end of treatment at 6 months.
  TNF-α measured from peripheral blood obtained via venipuncture using a bead-based multiplex assay (xMAP) with Luminex 200 flow cytometer. Unit of Measure: pg/mL.
C-Reactive Protein (CRP) | From enrollment to the end of treatment at 6 months.
  Measured in serum samples via immunonephelometry using a Dade Behring BNII nephelometer. Unit of Measure: mg/L.
Cognition: executive function | From enrollment to the end of treatment at 6 months.
  Executive function assessed using the computerized General Cognitive Assessment Battery (CAB) from CogniFit. The battery includes neuropsychological tests evaluating cognitive flexibility, divided attention, planning, visual and auditory perception, spatial perception, contextual memory, short-term visual and auditory memory, non-verbal memory, working memory, processing speed, naming, estimation, monitoring, response time, visual scanning, recognition, hand-eye coordination, focused attention, and inhibition. Test duration ranges from 25 to 45 minutes. Scores range from 0 to 800, with higher scores indicating better cognitive performance. Unit of Measure: CAB score (0-800).
Body Image perception | From enrollment to the end of treatment at 6 months.
  Body image perception assessed using the Spanish short version of the Multidimensional Body-Self Relations Questionnaire (MBSRQ). The questionnaire contains 45 items divided into two parts: General body image perception: scored on a Likert scale from 1 (Totally disagree) to 5 (Totally agree); and Satisfaction with specific body areas: scored on a Likert scale from 1 (Very dissatisfied) to 5 (Very satisfied). Higher scores indicate a more positive body image perception. Unit of Measure: points (Minimum Value: 45 - Maximum Value: 225).
3D and 4D Imaging | From enrollment to the end of treatment at 6 months.
  Morphological 4D images of participants were captured during each session using a 3D imaging system equipped with RGB-D devices. The 4D model represents morphological changes over time. Using cost-effective, wide-spectrum 3D acquisition technologies (RGB-D sensors), a 4D model was constructed as the core of a system for visualizing the human body over time. This model allows for precise and realistic visualization of body changes. Throughout the intervention, 3D morphological images of the participants were obtained, allowing them to observe their physical evolution through immersive Virtual Reality (VR)-a feature available only to the experimental group.

SECONDARY OUTCOMES:
Nutritional and Lifestyle measures: Physical Activity | From enrollment to the end of treatment at 6 months.
  Physical activity over the previous 7 days assessed using the International Physical Activity Questionnaire (IPAQ), Spanish Version, including 7 questions on frequency, duration, and intensity (vigorous and moderate), walking, and time spent sitting on a typical weekday. Higher scores indicate higher levels of physical activity. Unit of Measure: MET-minutes/week.
Nutritional and Lifestyle measures: Adherence to the Mediterranean Diet | From enrollment to the end of treatment at 6 months.
  Assessed using the 14-item PREDIMED Mediterranean Diet Adherence Questionnaire. Each item scores 0 or 1. Total scores range from 0 to 14, with scores ≥ 8 indicating good adherence and < 8 indicating low adherence to the Mediterranean Diet. Higher scores indicate better adherence. Unit of Measure: points (Minimum Value: 0 - Maximum Value: 14).
Nutritional and Lifestyle measures: Food Frequency Questionnaire | From enrollment to the end of treatment at 6 months.
  Dietary habits assessed using a 118-item Food Frequency Questionnaire adapted for the Spanish population. Scores range from 0 (never or <1/month) to 8 (+6 times per day). Higher scores indicate higher frequency of consumption of the specified food items. Unit of Measure: frequency (Minimum Value: 0 - Maximum Value: 8).
Nutritional and Lifestyle measures: 24-Hour Dietary Recall | From enrollment to the end of treatment at 6 months.
  Dietary intake assessed via three 24-hour dietary recalls (two weekdays and one weekend/holiday) to estimate nutrient and caloric intake. Higher values indicate higher intake. Unit of Measure: kilocalories (kcal) and grams of macronutrients per day.
Psychological measures: Premorbid Intelligence | From enrollment to the end of treatment at 6 months.
  Premorbid intelligence estimated based on the correct accentuation of 30 words, assessed using the Word Accentuation Test (TAP). The number of correct responses corresponds to an estimated IQ score based on the WAIS-IV scale. Higher scores indicate higher estimated premorbid intelligence. Unit of Measure: IQ points.
Psychological Measures: Emotional Eating | From enrollment to the end of treatment at 6 months.
  Assesses the influence of emotions on food choices through the Emotional Eater Questionnaire (CCE). 10 items scored on a Likert scale from 0 (Never) to 3 (Always). Higher scores indicate greater emotional influence on eating habits. Unit of Measure: points (Minimum Value: 0 - Maximum Value: 30).
Psychological Measures: Prefrontal Symptoms | From enrollment to the end of treatment at 6 months.
  Self-reported measure of cognitive, emotional, and behavioral disturbances in daily life, assessed using the Prefrontal Symptom Inventory, ISP-20 (Abbreviated Version). 20 items scored on a Likert scale from 0 (Never/almost never) to 4 (Always/almost always). Higher scores indicate more severe prefrontal symptoms. Unit of Measure: points (Minimum Value: 0 - Maximum Value: 80).
Psychological Measures: Impulsivity | From enrollment to the end of treatment at 6 months.
  Measures impulsivity across three subscales: cognitive (8 items), motor (10 items), and non-planning (12 items), assessed using the Barratt Impulsiveness Scale, BIS-11. Each item scored 0-4 (0=Rarely/Never, 4=Almost Always). Higher scores indicate greater impulsivity. Unit of Measure: points (Minimum Value: 0 - Maximum Value: 120).
Psychological Measures: Health-Related Quality of Life | From enrollment to the end of treatment at 6 months.
  Assesses physical and mental health-related quality of life using the Short Form-12 Health Survey (SF-12). 12 items scored from 0 (worst health) to 100 (best health). Higher scores indicate better health-related quality of life. Unit of Measure: points (Minimum Value: 0 - Maximum Value: 100).
Psychological Measures: Depression | From enrollment to the end of treatment at 6 months.
  21-item self-report questionnaire assessing depressive symptoms, measured using the Beck Depression Inventory-II (BDI-II). Items scored 0 (Not at all) to 3 (Severely). Higher scores indicate more severe depressive symptoms. Unit of Measure: points (Minimum Value: 0 - Maximum Value: 63).
Psychological Measures: Life Satisfaction | From enrollment to the end of treatment at 6 months.
  Measures global life satisfaction using the Satisfaction With Life Scale (SWLS). 5 items scored on a 7-point Likert scale (1=Completely disagree, 7=Completely agree). Higher scores indicate greater life satisfaction. Unit of Measure: points (Minimum Value: 5 - Maximum Value: 35).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Azorín López, Computer engineering, Principal Investigator — University of Alicante
Locations (1):
- University of Alicante, Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
At this time, the data cannot be shared because the patent registration process for the developed software is still ongoing. Until this stage is completed, it is not possible to consider sharing the Individual Participant Data (IPD) with other researchers. However, the project has been granted an extension and is currently in the analysis phase and in the process of creating a global database that integrates all the collected variables. Once this process is completed and the legal issues related to the patent are resolved, the data is expected to be published and made publicly available.

REFERENCES:
- [Background] González, Mariela. (2018). Validación del Cuestionario de Comedor Emocional (CCE) en Chile. Gen, 72(1), 21-24. Recuperado en 21 de noviembre de 2021, de http://ve.scielo.org/scielo.php?script=sci_arttext&pid=S001635032018000100005&lng=es&tlng=es.
- [Background] Martinez-Gonzalez MA, Fernandez-Jarne E, Serrano-Martinez M, Wright M, Gomez-Gracia E. Development of a short dietary intake questionnaire for the quantitative estimation of adherence to a cardioprotective Mediterranean diet. Eur J Clin Nutr. 2004 Nov;58(11):1550-2. doi: 10.1038/sj.ejcn.1602004. PMID 15162136
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Botella L, Corbella S, Belles L, Pacheco M, Maria Gomez A, Herrero O, Ribas E, Pedro N. Predictors of therapeutic outcome and process. Psychother Res. 2008 Sep;18(5):535-42. doi: 10.1080/10503300801982773. PMID 18816004
- [Background] Pons D, Atienza FL, Balaguer I, Garcia-Merita ML. Satisfaction with life scale: analysis of factorial invariance for adolescents and elderly persons. Percept Mot Skills. 2000 Aug;91(1):62-8. doi: 10.2466/pms.2000.91.1.62. PMID 11011872
- [Background] Rumbo-Rodriguez L, Sanchez-SanSegundo M, Ferrer-Cascales R, Garcia-D'Urso N, Hurtado-Sanchez JA, Zaragoza-Marti A. Comparison of Body Scanner and Manual Anthropometric Measurements of Body Shape: A Systematic Review. Int J Environ Res Public Health. 2021 Jun 8;18(12):6213. doi: 10.3390/ijerph18126213. PMID 34201258
- [Result] Zaragoza-Marti A, Sanchez-SanSegundo M, Ferrer-Cascales R, Gabaldon-Bravo EM, Laguna-Perez A, Rumbo-Rodriguez L. Effects of the Mediterranean Lifestyle During the COVID-19 Lockdown in Spain: Preliminary Study. Front Nutr. 2021 Jun 18;8:683261. doi: 10.3389/fnut.2021.683261. eCollection 2021. PMID 34222306
- [Result] N. García-D'urso, P. Climent-Pérez, M. Sánchez-Sansegundo, A. Zaragoza-Martí, A. Fuster-Guilló and J. Azorín-López, "A Non-Invasive Approach for Total Cholesterol Level Prediction Using Machine Learning," in IEEE Access, vol. 10, pp. 58566-58577, 2022, https://doi.org/10.1109/ACCESS.2022.3178419.
- [Result] Mauricio-Andres Zamora-Hernandez, Jose Andrez Chaves Ceciliano, Alonso Villalobos Granados, John Alejandro Castro Vargas, Jose Garcia-Rodriguez, Jorge Azorin-Lopez, "MDL+ a manufacturing description language to describe and control assembling tasks in industry 4.0", Logic Journal of the IGPL, 2022; jzac032, https://doi.org/10.1093/jigpal/jzac032
- [Result] L. F. Borja-Borja, J. Azorín-López, M. Saval-Calvo, A. Fuster-Guilló and M. Sebban, "Architecture for Automatic Recognition of Group Activities Using Local Motions and Context," in IEEE Access, vol. 10, pp. 79874-79889, 2022, https://doi.org/10.1109/ACCESS.2022.3195035
- [Result] Azorin-Lopez, Jorge, Fuster-Guilló, Andrés, Saval-Calvo, Marcelo, Villena Martínez, Víctor, Castillo Zaragoza, Juan Miguel, Garcia-d'Urso, Nahuel, Manchón Martínez, Cayetano, Ferrer-Cascales, Rosario, Zaragoza Martí, Ana, Sebban, Marc URI: http://hdl.handle.net/10045/119300
- See also: TECH4DIET webpage — https://tech4d.ua.es/en/home.html

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT07205029/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT07205029/ICF_001.pdf